CLINICAL TRIAL: NCT07051135
Title: HablaRÉ: Self-applied Online Training for Correcting Emotional Reasoning Biases in Public Speaking Anxiety. A Feasibility, Non-randomised Pilot Study.
Brief Title: HablaRÉ: Self-applied Online Training for Correcting Emotional Reasoning Biases in Public Speaking Anxiety.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Principal Investigator, Macarena Paredes Mealla, Principal investigator, Universitat Jaume I
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CEISH/86/2023-01
Record Dates: First submitted 2025-05-26; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Public Speaking Anxiety
Keywords: Emotional Reasoning; Public Speaking Anxiety; Anxiety; Emotional disorders; Feasibility; Internet intervention; Psychological treatment
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online treatment: Emotional Reasoning bias correction training (Experimental): Participants who meet the inclusion criteria will receive an Emotional Reasoning bias correction training called 'HablaRÉ' consisting of 10 self- administered sessions, delivered online with a duration of no more than 30 minutes each.
  Interventions: Device: "HablaRÉ": Emotional Reasoning bias correction training

INTERVENTIONS:
Device: "HablaRÉ": Emotional Reasoning bias correction training — The "HablaRÉ" bias correction training for Emotional Reasoning consists of ten online, self-administered sessions that last no more than 30 minutes each. These courses include practice tasks in addition to textual and audio-visual content. The explanation of ER bias, motivation to change, emotional psychoeducation, and the distinction between emotionally biassed and objective information are all addressed.

SUMMARY:
The project aims to assess the feasibility of self-administered training for individuals with public speaking anxiety, specifically targeting the reduction of emotional reasoning bias. It seeks to evaluate the interventions' usability, acceptability, satisfaction and adherence/compliance rates. In addition, the study intends to determine the feasibility of conducting a potential randomised clinical trial to evaluate the true impact of the intervention on emotional reasoning biases and public speaking anxiety levels.

DETAILED DESCRIPTION:
Public Speaking Anxiety (PSA), manifests as intense fear in public speaking or performance contexts, and while it is commonly seen in individuals with SAD, it can also occur independently. Studies show that 97% of individuals with SAD experience PSA, with approximately 40% suffering from severe PSA. PSA is associated with significant distress and detrimental effects on work, education, and social life. Several interventions, grounded in cognitive-behavioural principles, such as exposure therapies, have been proven effective in treating PSA, with both traditional and technology-based therapies demonstrating significant improvements in reducing anxiety and enhancing coping behaviours.

Despite the effectiveness of these treatments, relapse, non-improvement, or treatment discontinuation remain significant challenges. Comorbidity, affecting over 75% of individuals with affective disorders, worsens treatment outcomes and suggests the potential benefit of addressing transdiagnostic factors such as Emotional Reasoning (ER), a cognitive bias where individuals make judgements based on emotional responses rather than objective facts. Although ER has been targeted in interventions for spider phobia, no specific treatment for ER in PSA exists. The present study seeks to develop and assess the feasibility of "HablaRÉ" an intervention aimed at correcting ER biases in PSA patients. The study will evaluate the intervention's usability, acceptability, adherence, and its potential for a randomised clinical trial to determine its impact on ER bias and PSA levels.

A total of 30 participants will undergo training consisting of 10 self-administered daily sessions in which components such as psychoeducation on emotions and the detection of ER biases and their impact on behaviour.

ELIGIBILITY:
Inclusion Criteria:

1. Be of legal age.
2. Accept the informed consent.
3. Adequately understand/read Spanish.
4. Have access to a mobile device or computer with an Internet connection.
5. Not receiving any other psychological treatment for public speaking anxiety during the study period.
6. Have a score of 43 or higher on the Emotional reasoning scale (ERPSAS) AND/OR a score of 55 or higher on the Spanish version of the Public Speaking Anxiety Scale (PSAS-S) for fear of public speaking.
7. If taking prescribed medication for anxiety/depression, have had no changes in dosage for at least one month before the procedure.

Exclusion Criteria:

1. Not accepting the informed consent.
2. Being a minor.
3. Having a severe mental disorder (bipolar disorder, schizophrenia, or other psychotic disorders) or substance abuse (alcohol or other substances) or having active suicidal plans (suicide item in the ODSIS depression questionnaire ≥ 2) that would prevent participation in the program.
4. In the case of receiving medication, changes in medication during treatment will be evaluated but will not lead to exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Usability and acceptability | 2 evaluations: at post-treatment (just after treatment completion on the 10th day) and at 1-month follow up.
  The System Usability Scale (SUS) will be used to measure usability and acceptability (Brooke, 1996; Castilla et al., 2023). Patients rate their agreement with statements on a 5-point Likert scale (from 1, "Strongly Disagree", to 5, "Strongly Agree") as part of the SUS, which evaluates the usability of ICT applications using 10 items. The item values, which range from 0 to 4, are added up, and the total is multiplied by 2.5 to determine the overall score, which is expressed as a percentage (0-100). Better perceived usability are indicated by a larger percentage (Bangor et al., 2008).
Satisfaction with online training | 2 evaluations: at post-treatment (just after treatment completion on the 10th day) and at 1-month follow up.
  Using questions created by our team and previously used in technology-related studies, satisfaction with the intervention will be evaluated (Suso-Ribera, Castilla, Zaragozá, Ribera-Canudas, Botella, & García-Palacios, 2018). "To what extent are you satisfied with the app?" and "To what extent would you recommend the app?" are two examples of questions.
Adherence rates | 2 evaluations: at post-treatment (just after treatment completion on the 10th day) and at 1-month follow up.
  Adherence rates will be assessed according to the number of sessions completed by participants. Both the number of participants who fully complete the intervention (including the intervention, the final evaluation and the follow-up) and those who drop out will be considered. In these cases, it will be specifically identified at which stage of the process the drop-out occurred.
User interaction with the platform | 1 evaluation: at post-treatment (just after treatment completion on the 10th day).
  Interaction with the platform will be measured using access logs, specifically tracking the number of times participants log in for each session.

SECONDARY OUTCOMES:
Changes in ERPSAS Emotional Reasoning Public Speaking Anxiety Scale | 3 evaluations: at baseline before treatment onset, at treatment completion on the 10th day (Post-treatment evaluation) and 1-month follow up. Changes will be evaluated from pre-treatment to post-treatment and from post-treatment to 1 month follow-up.
  ERPSAS is a self-report instrument consisting of the presentation of 4 scenarios with different endings depending on whether objective safety or danger information is presented and whether there is an anxiety response or not. Based on these scenarios, the participant must measure, on a visual analogue scale (VAS) from 0 to 100, the degree of danger, safety, controllability, desire to avoid the situation and degree of discomfort. The sum of these scales provides a single perceived threat score, providing a measure to determine the presence of the emotional reasoning bias. If the participant evaluates emotional situations as threatening without objective information of danger, the presence of an Emotional Reasoning bias arises.
  The scale has a range of 0-96 points (M= 36.57; SD= 14.18). The higher the score, the greater the emotional reasoning bias, with the cut-off point being a score of 47. Participants scoring above half a standard deviation above the mean will be included.
Changes in Public Speaking Anxiety Scale | 3 evaluations: at baseline before treatment onset, at treatment completion on the 10th day (Post-treatment evaluation) and 1-month follow up. Changes will be evaluated from pre-treatment to post-treatment and from post-treatment to 1 month follow-up.
  The Public Speaking Anxiety Scale, which contains 17 items with a 5-point Likert-type response format (1=Not at all, 5=Extremely). This scale measures the presence and severity of cognitive, behavioural, and physiological symptomatology related to fear of public speaking, with a cut-off point of 73 (M= 49.33; SD= 12.88). Participants scoring above half a standard deviation above the mean will be included.
Changes in Overall Anxiety Severity and Impairment Scale | 3 evaluations: at baseline before treatment onset, at treatment completion on the 10th day (Post-treatment evaluation) and 1-month follow up. Changes will be evaluated from pre-treatment to post-treatment and from post-treatment to 1 month follow-up.
  OASIS is a 5-item self-report instrument that assesses a unidimensional factor related to the severity and frequency of anxiety symptoms, as well as behavioral avoidance and functional impairment associated with these symptoms in the past week. Each item has five response options, coded from 0 to 4. The total score is calculated by adding the values of all items, ranging from 0 to 20. Scores higher than 8 indicate the presence of anxiety symptoms. This scale has been validated online in a sample of patients with depression and anxiety, demonstrating good internal consistency (α=0.86), as well as adequate convergent and discriminantvalidities and sensitivity to change.
Changes in Overall Depression Severity and Impairment Scale | 3 evaluations: at baseline before treatment onset, at treatment completion on the 10th day (Post-treatment evaluation) and 1-month follow up. Changes will be evaluated from pre-treatment to post-treatment and from post-treatment to 1 month follow-up.
  ODSIS is a 5-item self-report instrument that the severity and functional impairment linked to depression over the past week. Each item has five response options coded from 0 to 4. The total score is calculated by summing the values of all items, ranging from 0 to 20. Scores of 5 or above suggest depressive symptoms. This scale was validated online using a sample of patients with depressive or anxiety disorders. It demonstrates excellent internal consistency (α=0.92), and its construct, convergent, and discriminant validities are supported.
Changes in Quality Life Index | 3 evaluations: at baseline before treatment onset, at treatment completion on the 10th day (Post-treatment evaluation) and 1-month follow up. Changes will be evaluated from pre-treatment to post-treatment and from post-treatment to 1 month follow-up.
  The QLI is a 10-item self-report instrument that assesses a single concept of quality of life across 10 dimensions using a ten-point Likert scale (1=poor; 10=excellent). The dimensions include physical well-being, psychological/emotional well-being, self-care and independent functioning, occupational functioning, interpersonal functioning, social-emotional support, community and services support, personal fulfilment, spiritual fulfilment, and overall perception of quality of life. The total score is the average of the item scores, ranging from 1 to 10 (1-4.5 = below average quality of life; 4.6-8.1 = average quality of life; 8.2-10 = above average quality of life). The QLI demonstrates high internal consistency (α=0.89) and test-retest reliability (0.89), with discriminant validity evidenced in a sample of psychiatric patients.
Reason for discontinuation of treatment | 1 evaluation: at post-treatment (until the end of the last session, up to 20 days)
  For participants who do not complete treatment, they will be asked voluntarily for the reason for discontinuing treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Macarena Paredes-Mealla, PhD Student, Principal Investigator — Universitat Jaume I; Carlos Suso-Ribera, PhD, Study Director — Universitat Jaume I; Azucena García Palacios, PhD, Study Director — Universitat Jaume I
Locations (1):
- University Jaume I, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lommen MJ, Engelhard IM, van den Hout MA, Arntz A. Reducing emotional reasoning: an experimental manipulation in individuals with fear of spiders. Cogn Emot. 2013;27(8):1504-12. doi: 10.1080/02699931.2013.795482. Epub 2013 May 16. PMID 23679871
- [Background] Arntz A, Rauner M, van den Hout M. "If I feel anxious, there must be danger": ex-consequentia reasoning in inferring danger in anxiety disorders. Behav Res Ther. 1995 Nov;33(8):917-25. doi: 10.1016/0005-7967(95)00032-s. PMID 7487851
- [Background] Paredes-Mealla M, Martinez-Borba V, Miragall M, Garcia-Palacios A, Banos RM, Suso-Ribera C. Is there evidence that emotional reasoning processing underlies emotional disorders in adults? A systematic review. Curr Psychol. 2022 Nov 9:1-17. doi: 10.1007/s12144-022-03884-4. Online ahead of print. PMID 36406838